CLINICAL TRIAL: NCT04086459
Title: PET/MRI Study on the Neurological Mechanism of rTMS Treatment for Heroin Addiction by Stimulating Left Dorsolateral Prefrontal Cortex
Brief Title: PET/MRI Study on the Neurological Mechanism of rTMS Treatment for Heroin Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Addiction-No.1
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Heroin Addiction; Relapse
Keywords: Repetitive transcranial magnetic stimulation; Functional magnetic resonance imaging; Positron emission tomography
MeSH Terms: conditions — Heroin Dependence; Recurrence | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Three groups (two groups of heroin addiction during methadone maintenance treatment and one healthy control group) were included in this study design. One heroin addiction group was administered active repetitive transcranial magnetic stimulation (rTMS) while another heroin addiction group was administered sham. The healthy control group was not given rTMS, just as control.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Either the participants, care providers, or outcomes assessors did not know which repetitive transcranial magnetic stimulation is active or sham.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active repetitive transcranial magnetic stimulation (Active Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham repetitive transcranial magnetic stimulation (Sham Comparator)
  Interventions: Device: Repetitive transcranial magnetic stimulation
- No repetitive transcranial magnetic stimulation (No Intervention)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Those receiving experimental treatment will receive 20 sessions of rTMS, stimulation protocol included 20 sessions within 30 days (once a day, 5 days/week, 4 weeks, 10 Hz frequency, pulse intensity 100% of the resting motor threshold, 50 pulses per train, inter train pause of 10 s, 40 stimulation trains, 2000 pulses/ session)
  Arms: Active repetitive transcranial magnetic stimulation; Sham repetitive transcranial magnetic stimulation

SUMMARY:
Heroin addiction is a serious problem and the relapse rate of existing treatment methods is extremely high. Recently, international journals such as Science reported that repetitive transcranial magnetic stimulation (rTMS) can reduce the craving of addicts, alleviate depression and anxiety symptoms, and is expected to become an effective treatment. Our preliminary experiment using rTMS to stimulate the left dorsolateral prefrontal cortex of heroin addicts also showed similar effects, however, the mechanism is unclear. Previously, the investigators found that the functional connectivity between left executive control network and default mode network was negatively correlated relapse behavior, while the functional connectivity between salience network and default mode network was positively correlated with relapse behavior. Studies have shown that dopamine dysfunction in addicts and brain metabolism is the biological basis of network connectivity. It suggests that elucidating the relationship between the characteristics of large brain network connectivity and the level of dopamine receptor and relapse behavior in addicts is hopeful to further understand the neurological mechanism of rTMS treatment for addiction. In this project, the investigators intend to observe the changes of brain network connectivity, glucose metabolism and dopamine D2 receptor before and after rTMS treatment in addicts from the perspective of large brain network by combining PET/MRI with psychobehavioral approach. The relationship between rTMS and relapse behavior will be deeply analyzed to provide scientific basis for the development of effective treatment programs.

ELIGIBILITY:
Inclusion Criteria for Heroin-dependent Participants:

* Clinical diagnosis of heroin addiction
* Have been receiving treatment in a methadone maintenance treatment program for no less than 6 months
* have been on a stable dose for at least 1 month before entering the study
* Right-handed

Inclusion Criteria for Healthy Control Participants:

* Clinical diagnosis of Healthy Control
* Right-handed

Exclusion Criteria for all Participants:

* Current or past psychiatric illness other than heroin and nicotine dependence
* Neurological signs and/or history of neurological disease
* History of head trauma
* History of cardiovascular or endocrine disease
* Current medical illness or recent medicine use
* Presence of magnetically active objects in the body
* Claustrophobia or any other medical condition that would preclude the participant from lying in the PET/MRI scanner for approximately 40 min.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of craving | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Craving scores will be assessed with visual analogue scale
Change of protracted-abstinence symptoms | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Protracted-abstinence symptoms scores will be assessed with protracted symptoms questionnaire
Change of depress symptoms | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Depress symptoms scores will be assessed with Beck Depression Inventory
Change of anxiety symptoms | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Anxiety symptoms scores will be assessed with Hamilton Anxiety Scale
Change of impulsive behaviors | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Impulsive behaviors scores will be assessed with Barratt impulsiveness scale
Change of sleep | Baseline, 1 week later, 1,2,3,4,5,6 months later
  Sleep scores will be assessed with Pittsburgh sleep quality index
Change of functional connectivity between dorsolateral prefrontal cortex and whole brain | Baseline, 1 week later, 1,3,6 months later
  Functional connectivity based on dorsolateral prefrontal cortex will be measured with magnetic resonance imaging based on blood oxygen level dependence
Change of gray matter volume of whole brain | Baseline, 1 week later, 1,3,6 months later
  Gray matter volume will be measured with magnetic resonance imaging (high resolution T1-weighted image)
Change of white matter integrity of whole brain | Baseline, 1 week later, 1,3,6 months later
  Fractional anisotropy, axial diffusivity and radial diffusivity will be measured with magnetic resonance imaging (diffusion tensor imaging)
Change of availability of dopamine 2 receptor of whole brain | Baseline, 1 month later
  Accumulation of 11C-raclopride will be analyzed by time-related Positron emission tomography
Change of metabolism of glucose in the brain | Baseline, 1 month later
  Accumulation of 18F-FDG will be analyzed by time-related Positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Longxiao Wei, phd, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No